CLINICAL TRIAL: NCT04721080
Title: Effects of Pulmonary Tuberculosis Sequelae on Functional Outcomes in Patients With COPD
Brief Title: Pulmonary Tuberculosis Sequelae in Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: IKC145
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Copd; Tuberculosis; Quality of Life
Keywords: copd; tuberculosis; exercise capacity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients with tuberculous sequelae: COPD patients with tuberculous sequelae
  Interventions: Other: Functional Outcome Measurements
- COPD patients without tuberculosis sequela: COPD patients with tuberculous sequelae
  Interventions: Other: Functional Outcome Measurements

INTERVENTIONS:
Other: Functional Outcome Measurements — Dyspnea Exercise capacity Quality of life assessment

SUMMARY:
It is known that there is a complex relationship between tuberculosis and COPD. Post-tuberculosis airway disease or COPD associated with tuberculosis occurs in a significant portion of tuberculosis patients. However, it was observed that mortality rates and exacerbation rates of COPD patients with tuberculosis sequel were higher. However, the effect of tuberculosis sequela on functional outcomes in COPD patients has not been investigated in the studies.

The aim of this study is to determine whether the previous tuberculosis sequelae has a functional effect on patients with COPD.

DETAILED DESCRIPTION:
This research is planned as a cross-sectional study. It will start within one week following the approval of the ethics committee and will be completed within one year. The universe of the study is S.B.Ü. Dr. Suat Seren Chest Diseases and Surgery Training and Research Hospital consists of patients who apply to Pulmonary Rehabilitation Outpatient Clinic. Participants will consist of two different groups: COPD patients with tuberculosis and COPD patients without tuberculosis. The voluntary principle will be taken into account in participating in the research.

Within the scope of the evaluation; Demographic and clinical information of the people who will participate in the study will be recorded, and Thorax CT and PFT examinations performed within the polyclinic service within the last 1 month will be evaluated. Saint George Respiratory Questionaire (SGRQ), 6-minute walk test (6MWT), Medical Research Council Dyspnea Scale (MRC), COPD assessment test (CAT) will be applied to the patients. Regarding the illness histories, the number of hospitalizations and emergency admissions in the last 1 year will be recorded. Detailed tuberculosis anamneses will also be taken from patients with tuberculosis sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being over 18 years old
* Having thorax CT in the last 1 month
* Having PFT examination performed in the last 1 month

Exclusion Criteria:

* Being in a COPD attack
* The patient has additional pulmonary comorbidity such as Lung Ca, bronchiectasis, lung fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with tuberculous sequelae and COPD patients without tuberculosis sequela
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | 6 minutes- baseline
  Six minutes walk test

SECONDARY OUTCOMES:
Dyspnea Assessment | 5 minutes- baseline
  Medical Research Council Scale(MRC)
COPD Assessment | 5 minutes- baseline
  COPD Assessment Test (CAT
Quality of Life Assessment | 20 minutes- baseline
  St. George Respiratory Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Sahin, Principal Investigator — Izmir Dr. Suat Seren Chest Diseases and Surgery Training and Research Hospital
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)